CLINICAL TRIAL: NCT03449654
Title: Effect of Liraglutide on Vascular Inflammation in Type-2 Diabetes: A Randomized, Placebo-controlled, Double-blind, Parallel Clinical PET/CT Trial The Liraflame Trial
Brief Title: Effect of Liraglutide on Vascular Inflammation in Type-2 Diabetes
Acronym: LIRAFLAME
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Steno Diabetes Center Copenhagen (Other)
Collaborators: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Peter Rossing, MD, chief phycisian, Dr. Med., Steno Diabetes Center Copenhagen
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: H-16044546
Record Dates: First submitted 2017-12-07; First posted 2018-02-28 (Actual); Last update posted 2020-06-11 (Actual); Status verified 2020-06

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Liraglutide

STUDY DESIGN:
Intervention Model Description: Randomized, Placebo-controlled, Parallel
Who Masked: Participant, Investigator
Masking Description: Dobbelt-blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Liraglutide (Other)
  Interventions: Drug: Liraglutide
- placebo (Other)
  Interventions: Drug: Placebo (for liraglutide)

INTERVENTIONS:
Drug: Liraglutide — Liraglutid
  Arms: Liraglutide
Drug: Placebo (for liraglutide) — Placebo (for liraglutide)
  Arms: placebo

SUMMARY:
The objective of this study is to evaluate the mechanism behind the anti-atherogenic effects of liraglutide.

In a randomized, placebo-controlled, double-blind, parallel trial we will included 100 patients with type 2 diabetes. Patients will be randomized 1:1 to an active treatment period of 26 weeks or placebo for 26 weeks.

The primary endpoint is change from baseline to week 26 in vascular inflammation, assessed by Flour Deoxy Glucose (FDG)-Positron Emission Tomography/Computed Tomography (PET/CT)

DETAILED DESCRIPTION:
Despite multifactorial treatment patients with type 2 diabetes are still at high risk of cardiovascular disease. The clinical LEADER trial demonstrated a reduction in cardiovascular events in patients with type 2 diabetes treated with the GLP-1 receptor agonist liraglutide and there are a number of studies indicating that liraglutide has a positive effect on the vascular phenotype. Several of the animal or ex vivo studies suggest an anti-inflammatory mechanism behind this effect. However, no in vivo human studies have been undertaken to test this hypothesis and it would be of significance to determine the precise mechanism since atherosclerosis has large prognostic impact in patients with type 2 diabetes.

The objective of this study is to evaluate the mechanism behind the anti-atherogenic effects of liraglutide.

In a randomized, placebo-controlled, double-blind, parallel trial we will included 100 patients with type 2 diabetes. Patients will be randomized 1:1 to an active treatment period of 26 weeks or placebo for 26 weeks.

The primary endpoint is change from baseline to week 26 in vascular inflammation, assessed by Flour Deoxy Glucose (FDG)-Positron Emission Tomography/Computed Tomography (PET/CT). FDG-PET/CT is currently the only clinically available technique for specific in vivo evaluation of vascular inflammation and for quantification of the effects of medical intervention on plaque inflammation. FDG-PET of arteries has been proven very reproducible and therefore has high power to show a treatment effect in a smaller group of patients.

A number of complementary methods exist that assess different steps in the atherogenesis like endothelial function (e.g. endo-PAT, glycocalyx measurement), artery wall thickening (e.g. carotid intima media thickness), or coronary atherosclerosis (e.g. coronary artery calcium score). For comparison these other methods will be included as secondary endpoints as they are generally more accessible and less expensive.

ELIGIBILITY:
Inclusion Criteria:

1. Given written informed consent
2. Male or female patients >50 years with type 2 diabetes (WHO criteria)
3. HbA1c ≥ 48 mmol/mol (6.5 %)
4. eGFR ≥ 30 ml/min/1.73 m2 (estimated by CKD-epi formula)
5. Stable glucose-lowering medication (excluding oral glucocorticoids, calcineurin inhibitors, dipeptidyl peptidase 4 (DPP4) inhibitors, glucagon like peptide-1 agonists and other agents, which in the investigator's opinion could interfere with the effect of liraglutide)for at least 4 weeks before the baseline PET/CT
6. Stable/no treatment of hypercholesterolemia 4 weeks before baseline PET/CT
7. Must be able to communicate with the investigator and understand informed consent.

Exclusion Criteria:

1. Type 1 diabetes mellitus
2. Chronic pancreatitis / previous acute pancreatitis
3. Known or suspected hypersensitivity to trial product(s) or related products
4. Treatment 90 days prior to screening with oral glucocorticoids, calcineurin inhibitors, dipeptidyl peptidase 4 (DPP4) inhibitors, glucagon like peptide-1 agonists and other agents, which in the investigator's opinion could interfere with the effect of liraglutide
5. Cancer or any other clinically significant disorder, except for conditions associated with type 2 diabetes history, which in the investigators opinion could interfere with the results of the trial
6. Clinical signs of diabetic gastroparesis
7. Previous bowel resection
8. Impaired liver function (transaminases > two times upper reference levels)
9. Inflammatory bowel disease
10. Weight >150 kg
11. Females of childbearing potential who are pregnant, breast-feeding, intend to become pregnant or are not using adequate contraceptive methods
12. Known or suspected abuse of alcohol or narcotics
13. Subjects with personal or family history of medullary thyroid carcinoma or a personal history of multiple endocrine neoplasia type 2

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2017-10-26 (Actual); Primary Completion 2019-08-16 (Actual); Study Completion 2019-08-16 (Actual)

PRIMARY OUTCOMES:
Change in vascular inflammation | baseline to week 26
  Change in vascular inflammation assessed by FDG PET/CT

SECONDARY OUTCOMES:
Change in Endothelial dysfunction | baseline to week 26
  Change in endothelial dysfunction assessed with endo-PAT
Change in Endothelial dysfunction | baseline to week 13 and 26
  Change in endothelial dysfunction, assessed as sublingual glycocalyx measurement
Coronary artery calcium score | baseline to week 26
  Change coronary artery calcium score (absolute values)
Carotid intima media thickness | baseline to week 26
  Change in carotid intima media thickness measured by ultrasound

OTHER OUTCOMES:
Autonomic nervous system function | baseline to week 26
  Change in cardiovascular autonomic neuropathy indices

CONTACTS AND LOCATIONS:
Locations (1):
- Steno Diabetes Center Copenhagen, Gentofte Municipality, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wretlind A, Curovic VR, de Zawadzki A, Suvitaival T, Xu J, Zobel EH, von Scholten BJ, Ripa RS, Kjaer A, Hansen TW, Vilsboll T, Vestergaard H, Rossing P, Legido-Quigley C. Ceramides are decreased after liraglutide treatment in people with type 2 diabetes: a post hoc analysis of two randomized clinical trials. Lipids Health Dis. 2023 Sep 26;22(1):160. doi: 10.1186/s12944-023-01922-z. PMID 37752566
- [Derived] Wretlind A, Zobel EH, de Zawadzki A, Ripa RS, Curovic VR, von Scholten BJ, Mattila IM, Hansen TW, Kjaer A, Vestergaard H, Rossing P, Legido-Quigley C. Liraglutide Lowers Palmitoleate Levels in Type 2 Diabetes. A Post Hoc Analysis of the LIRAFLAME Randomized Placebo-Controlled Trial. Front Clin Diabetes Healthc. 2022 Mar 4;3:856485. doi: 10.3389/fcdhc.2022.856485. eCollection 2022. PMID 36992761
- [Derived] Zobel EH, Wretlind A, Ripa RS, Rotbain Curovic V, von Scholten BJ, Suvitaival T, Hansen TW, Kjaer A, Legido-Quigley C, Rossing P. Ceramides and phospholipids are downregulated with liraglutide treatment: results from the LiraFlame randomized controlled trial. BMJ Open Diabetes Res Care. 2021 Sep;9(1):e002395. doi: 10.1136/bmjdrc-2021-002395. PMID 34518158
- [Derived] Ripa RS, Zobel EH, von Scholten BJ, Jensen JK, Binderup T, Diaz LJ, Curovic VR, Hansen TW, Rossing P, Kjaer A. Effect of Liraglutide on Arterial Inflammation Assessed as [18F]FDG Uptake in Patients With Type 2 Diabetes: A Randomized, Double-Blind, Placebo-Controlled Trial. Circ Cardiovasc Imaging. 2021 Jul;14(7):e012174. doi: 10.1161/CIRCIMAGING.120.012174. Epub 2021 Jun 30. PMID 34187185